CLINICAL TRIAL: NCT04676581
Title: Risk Benefit Ratio of Hirudotherapy: Retrospective Single-center Study of 37 Cases Over a Period of 9 Years
Acronym: AMLEE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0136
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Leeches; Healthcare Associated Infection
Keywords: Leeches; Healthcare-associated infection; Hirudo Medicinalis
MeSH Terms: conditions — Cross Infection | interventions — Leeching

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aeromonas infection
  Interventions: Other: Leech Therapy
- No infected
  Interventions: Other: Leech Therapy
- bacterial infection
  Interventions: Other: Leech Therapy

INTERVENTIONS:
Other: Leech Therapy — Patient who received leeches (for more than 2 days) at the Amiens University Hospital over a period of 9 years (2010-2018)

SUMMARY:
Venous congestion in transplanted or re-implanted tissues remains a common and chal-lenging complication in plastic and reconstructive surgery. Local application of medicinal leeches is effective to reduce postoperative venous congestion of the flap and to restore normal blood flow. However, leech therapy is associated with a number of risks, including infections. Indeed, leeches maintain a symbiotic relationship with Aeromonas species in order to digest blood in their gut. Aeromonas spp. infections can occur 1 to 30 days post-application of leeches and are associated with a dramatic decrease in flap salvage rates (88 to 30%). For these reasons, prophylactic antibiotics and, external decontamination are widely recommended throughout the course of leech therapy.

The aim of this study is to investigate the prevalence of side effects (anemia and infection) from patients treated with leeches in French Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received leeches (for more than 2 days) at the Amiens University Hospital over a period of 9 years (2010-2018)

Exclusion Criteria:

* Hirudotherapy outside the inclusion period
* Hirudotherapy or less than 2 days of treatment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who received leeches (for more than 2 days) at the Amiens University Hospital over a period of 9 years (2010-2018)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
number of patients requiring a second surgery | 9 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No